CLINICAL TRIAL: NCT06072079
Title: Studies of Structural Chromosome Rearrangements to Identify Genes Involved in Congenital Brain Disorders
Brief Title: Structural Chromosome Rearrangements and Brain Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Lindstrand, MD, PhD; Adjunct Professor, Karolinska Institutet
Other Study IDs: 2019-02078
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Rare Diseases; Genetic Disease; Chromosome Abnormality
Keywords: genome sequencing; structural variants
MeSH Terms: conditions — Rare Diseases; Genetic Diseases, Inborn; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The project is focused on the detailed study of structural genomic variants (SVs). Such genetic mutations are in fact alterations in the DNA molecule structure and include copy number variants, inversions and translocations. A single event may affect many genes as well as regulatory regions and the specific phenotypic consequences will depend on the location, genetic content and type of SV. Many times, the specific disease-causing mechanism is not known. Here, the plan is to study the molecular genetic behavior of structural variants as well as the underlying mutational mechanisms involved.

First, genome sequencing will be done to pinpoint the chromosomal breakpoints at the nucleotide level, characterize the genomic architecture at the breakpoints and study the relationship between structural variants and SNVs. Second, the aim is to study how structural variants impact gene expression. Finally, disease mechanisms will be functionally explored in vivo using zebrafish and in vitro using primary patient cells and induced pluripotent stem cells.

The studies will focus on the origin, structure and impact of structural variation on human disease. The results will directly lead to a higher mutation detection rate in genetic diagnostics. Through a better understanding of disease mechanisms the findings will also assist in the development of novel biomarkers and therapeutic strategies for patients with rare genetic disorders.

DETAILED DESCRIPTION:
PROJECT DESCRIPTION Aim 1) What are the molecular mechanisms of formation for structural genomic variants?

There is already WGS data from more than 500 individual SVs. To understand underlying mutational and disease mechanisms, structural variant detection will be combined with positional information for the rearrangement. This will be particularly important for duplications (the location of the duplicated genomic segment is key to a correct clinical interpretation) and for complex rearrangements. Second, the exact breakpoint will be established and breakpoint junctions analyzed for sequence motifs.

Aim 2) What are the molecular mechanisms involved in disease pathology?

First WGS will be used to identify and characterize structural variants. Next, to understand how the candidate disease gene(s) affected by the SVs cause clinical symptoms, the cellular mechanisms involved in disease pathology will be studied in three ways:

Part 1. In vitro studies of primary cells: Effects on expression and splicing, will be evaluated in patient cells (fibroblasts or B cell lines) with RT-PCR, qPCR and Western blot.

Part 2. In vitro studies in patient-derived models: In selected cases, induced-pluripotent stem cells and neural progenitor cells (NES cells) will be generated, which will provide an opportunity to directly study the effects of early neurogenesis in cells from the patient and compare to cells derived from normal controls. The investigators are interested in studying both early neurogenesis in 2D culture using the NES cells, as well as generating another developmentally relevant model, brain organoids (mini brains), in 3D culture directly from iPS cell lines. Organoid 3D culture recapitulates development of various brain regions and is therefore a unique tool to investigate brain disorders. Furthermore, the 3D neural culture could improve cell maturity and stimulate expression of disease phenotypes that facilitate better understanding the disease mechanisms.

Part 3. In vivo studies in a zebrafish model: Zebrafish (Danio rerio) is a well-functioning in vivo system for studies of normal and abnormal embryological development. Duplications are simulated by RNA overexpression and deletion through CRISPR/Cas9 induced gene disruption or morpholino knock down. Assessment of the phenotypes is designed in accordance with the those observed in patients (e.g. head size, craniofacial defects, cardiovascular malformations, cilia defects).

Aim 3) How does structural genomic variants impact gene expression?

Long range effects will be studied in three ways. Part 1. To assess the clinical impact of TAD disruptions, CNV data from the Clinical Genetics array database (data from over 6200 children with rare NDDs), LocusDB SV (SV calls from >1000 patients with rare diseases analyzed by WGS at Clinical Genomics SciLifeLab) and publicly available databases (DECIPHER, ICCG and SWEGEN) will be analysed. The Bioinformatic analysis will combine information on phenotypic overlap between known-disease genes surrounding the SV and the patients' characteristics, as well as on physical overlap with tissue-specific enhancers and TAD regions. Novel computational approaches will be designed for the discovery of genes disrupted by similar mechanisms. Follow-up studies will involve further patient characterization and customized RNA studies.

Part 2. Transcriptome analysis of patient samples is done by RNA-seq. Since not every gene is transcriptionally active in every cell, a key to successfully achieving this aim is access to biologically relevant samples. Often biopsies are not available therefore, in those cases, iPS cells are an alternative way to study biologically relevant effects on RNA expression. In cases with paired WGS and RNA-seq data, we will integrate changes in transcription levels and ASE as a readout for the SVs effect on neighboring genes.

Part 3. Cell and animal studies: Introduction of specific SVs with CRISPR/Cas9 in human cell lines will be done when the primary cells are unavailable and zebrafish lines created under goal 2 may also be used to evaluate global effects of SVs on an organism level.

ELIGIBILITY:
Inclusion Criteria:

Individual with a suspected rare disease and/or chromosomal abnormality

Exclusion Criteria:

No suspected rare disease or chromosome abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals that have undergone genetic investigations due to a suspected rare disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Understanding disease mechanisms | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Lindstrand, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided